CLINICAL TRIAL: NCT01312883
Title: Center for Achieving and Sustaining Improved Health in Harlem: Patient Education to Reduce Postpartum Depressive Symptoms Among Minority Women
Brief Title: Mothers Avoiding Depression Through Empowerment Intervention Trial
Acronym: MADE IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Elizabeth A. Howell, MD, MPP, Mount Sinai School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2P60MD000270-06 (NIH); P60MD000270 (NIH)
Record Dates: First submitted 2011-03-08; First posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as usual (No Intervention): Participants will receive standard postpartum education and discharge materials provided by the hospital and a list of community and Internet resources by mail.
- Behavioral education (Experimental): Participants will receive behavioral education on postpartum depression and a list of community and Internet resources by mail.
  Interventions: Behavioral: Behavioral education intervention

INTERVENTIONS:
Behavioral: Behavioral education intervention — One education session with a social worker while at the hospital, provision of an educational pamphlet and summary sheet for partner, a needs assessment by the social worker 2 weeks after hospital discharge, and additional patient education and reinforcement of self-management skills, as needed
  Arms: Behavioral education

SUMMARY:
Postpartum depressive symptoms are a major health problem that affects hundreds of women annually. The investgators propose to test an intervention to reduce postpartum depressive symptoms and prevent elevated levels of depressive symptoms in postpartum mothers by preparing and educating women about specific situational triggers of depressive symptoms, by bolstering personal and social resources, by enhancing self-management skills to buffer postpartum demands, and by increasing access to existing healthcare and community resources available to postpartum mothers.

DETAILED DESCRIPTION:
Postpartum depression (PPD) is a disorder affecting many women after delivery of a child. Up to 50% of mothers may experience some depressive symptoms after giving birth, and up to 25% of them will develop major depressive disorder. Some situational factors that place mothers at risk of PPD may be changed or minimized, including social support, the mother's efficiency in handling situational stress, and distress from physical symptoms. Preparing mothers to identify potential situational triggers of depressive symptoms, enhancing their postpartum self-management skills , and providing them access to the proper social and healthcare resources may prevent them from developing major depression. This study will test the efficacy of a brief intervention that aims to prevent PPD by preparing mothers to deal with stressful triggers and depressive symptoms.

This study will last 6 months. Participants will be randomly assigned to receive either treatment as usual or the behavioral education intervention. The intervention will involve two parts. First, after giving birth and while still in the hospital, participants will complete an education session with a social worker and receive written materials about PPD. Then, 2 weeks after discharge from the hospital, participants will receive a call from the social worker, who will conduct a needs assessment that addresses participants' physical and emotional health. If a participant is experiencing distress, the social worker will refer her to appropriate resources and will reinforce self-management skills. All participants will receive a list of community and hospital resources by mail.

Study assessments will take place at 3 weeks, 3 months, and 6 months after study entry. At these points, participants will complete a 20-minute survey with a research assistant about their health, mood, and basic demographic information.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the Maternity Unit at Mount Sinai Hospital
* Infant has a birth weight greater than or equal to 2,500 grams
* Infant has a 5-minute Apgar score greater than or equal to 7
* Self-identifies as Black/African American or Hispanic/Latina; White or minority other than Black/African American or Hispanic/Latina will be referred to a parallel study with the same protocol at Mount Sinai Hospital
* Speaks English or Spanish
* Has a working telephone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2007-09; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is to evaluate the effectiveness in a randomized controlled trial of a patient education intervention to reduce depressive symptoms among Black and Hispanic postpartum women. | Measured at baseline
The primary outcome measure is to evaluate the effectiveness in a randomized controlled trial of a patient education intervention to reduce depressive symptoms among Black and Hispanic postpartum women. | Measured at 3 weeks postpartum
The primary outcome measure is to evaluate the effectiveness in a randomized controlled trial of a patient education intervention to reduce depressive symptoms among Black and Hispanic postpartum women. | Measured at 3 months postpartum
The primary outcome measure is to evaluate the effectiveness in a randomized controlled trial of a patient education intervention to reduce depressive symptoms among Black and Hispanic postpartum women. | Measured at 6 months postpartum

SECONDARY OUTCOMES:
Breastfeeding continuation rate and Physical functioning | Measured at baseline and after 3 weeks, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Howell, MD, MPP, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

REFERENCES:
- [Derived] Bodnar-Deren S, Klipstein K, Fersh M, Shemesh E, Howell EA. Suicidal Ideation During the Postpartum Period. J Womens Health (Larchmt). 2016 Dec;25(12):1219-1224. doi: 10.1089/jwh.2015.5346. Epub 2016 May 26. PMID 27227751
- [Derived] Balbierz A, Bodnar-Deren S, Wang JJ, Howell EA. Maternal depressive symptoms and parenting practices 3-months postpartum. Matern Child Health J. 2015 Jun;19(6):1212-9. doi: 10.1007/s10995-014-1625-6. PMID 25374288
- [Derived] Howell EA, Bodnar-Deren S, Balbierz A, Parides M, Bickell N. An intervention to extend breastfeeding among black and Latina mothers after delivery. Am J Obstet Gynecol. 2014 Mar;210(3):239.e1-5. doi: 10.1016/j.ajog.2013.11.028. Epub 2013 Nov 18. PMID 24262719
- [Derived] Negron R, Martin A, Almog M, Balbierz A, Howell EA. Social support during the postpartum period: mothers' views on needs, expectations, and mobilization of support. Matern Child Health J. 2013 May;17(4):616-23. doi: 10.1007/s10995-012-1037-4. PMID 22581378
- [Derived] Howell EA, Balbierz A, Wang J, Parides M, Zlotnick C, Leventhal H. Reducing postpartum depressive symptoms among black and Latina mothers: a randomized controlled trial. Obstet Gynecol. 2012 May;119(5):942-9. doi: 10.1097/AOG.0b013e318250ba48. PMID 22488220